CLINICAL TRIAL: NCT02679651
Title: Diagnostic Modeling for Pedal Fat Pad Atrophy
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jeffrey A. Gusenoff, MD, Associate Professor, University of Pittsburgh
Other Study IDs: PRO15060610
Record Dates: First submitted 2016-02-06; First posted 2016-02-10 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Fat Pad Atrophy; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control group: Healthy Adults without foot pain
  Interventions: Other: Ultrasound of the foot; Other: Pedobarograph Measurements; Other: Manchester Foot Pain and Disability Index
- DIsease group: Adults diagnosed with fat pat atrophy and report symptoms of foot pain and have participated in clinical trial to treat fat pad atrophy.
  Interventions: Other: Ultrasound of the foot; Other: Pedobarograph Measurements; Other: Manchester Foot Pain and Disability Index

INTERVENTIONS:
Other: Ultrasound of the foot — An ultrasound will be used to determine the thickness of the fat pad
Other: Pedobarograph Measurements — This non-invasive device measures the force and pressure of the foot while standing and walking.
Other: Manchester Foot Pain and Disability Index — This is a patient completed questionnaire that assesses level of function from the past month specific to foot pain.

SUMMARY:
The investigators hypothesize that there is a difference in plantar tissue thickness, plantar pressure, and pain score in patients diagnosed with plantar fat pad atrophy compared to healthy, foot-type matched controls. Results will be measured objectively using ultrasound for tissue thickness, optical pedobarograph for plantar pressure, and Manchester foot pain and disability index (MFPDI) for pain score. Furthermore, investigators predict that these results will help establish criteria for fad pad atrophy diagnosis in the clinic as well as determine which patients would receive greatest benefit from fat grafting to the foot.

DETAILED DESCRIPTION:
Human feet must bear the entire weight of the body. Feet have fat pads on their plantar surface that act as shock absorbers between the skin and bone. However, repetitive mechanical stress throughout a person's lifetime leads to gradual atrophy of these fat pads. In addition to this age-related degeneration, fat pad atrophy can be caused by other mechanisms such as abnormal foot mechanics, steroid use, and collagen vascular disease. Regardless of the cause, many patients with plantar fat pad atrophy experience considerable pain and loss of function.

Previous studies have negatively correlated plantar soft tissue thickness with plantar pressure, with the loss of plantar fat being a fundamental mechanism associated with pressure-related foot disorders. Increased pressure from fat pad atrophy is commonly managed with padded socks, insoles, and shoe modification. However, these extrinsic strategies are totally dependent on patient compliance, and devices must be replaced as soon as they begin to break down. Another treatment option includes silicone injections into the plantar aspect of the foot. In one study, patients receiving silicone treatment experienced increased plantar tissue thickness and decreased plantar pressure, but these cushioning properties decreased over time and the need for additional booster injections was ultimately suggested. Furthermore, silicone has been known to migrate away from the injection site and has been found in the inguinal lymph nodes of patients.

A different strategy that is gaining momentum is autologous fat grafting to the foot. Taking a patient's own tissue, often from the abdomen or thigh, and transplanting it to areas of plantar fat pad atrophy may reduce pressure in a more natural and permanent manner. Only one study to date has been published on autologous fat grafting to the foot, but the patients were receiving concurrent surgical procedures with their fat grafting and the results were reported subjectively by the patients.

In this study, the investigators hypothesize that there is a difference in plantar tissue thickness, plantar pressure, and pain score in patients diagnosed with plantar fat pad atrophy compared to healthy, foot-type matched controls. Results will be measured objectively using ultrasound for tissue thickness, optical pedobarograph for plantar pressure, and Manchester foot pain and disability index (MFPDI) for pain score. Furthermore, the investigators predict that these results will help establish criteria for fad pad atrophy diagnosis in the clinic as well as determine which patients would receive greatest benefit from fat grafting to the foot.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Patients without foot pain at the plantar surface of the foot near the head of the metatarsals
3. 6 months post any surgical intervention to the foot
4. Subjects must be determined by the PI or a Co-Investigator to not suffer from pedal pad atrophy

Exclusion Criteria:

1. Age less than 18 years
2. Inability to provide informed consent
3. Feet with open ulcerations or osteomyelitis
4. Diabetics: Type I and II
5. Active infection anywhere in the body
6. Diagnosed with cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment
7. Pregnancy
8. Tobacco use: Last use within 1 year per patient report

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 healthy, age matched adults with normal foot fat pads to compare to 30 patients in the fat pad atrophy group from our other IRB approved clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Plantar fat pad thickness | Screening
  Fat pad thickness measured via ultrasound
Plantar foot pressure | Screening
  Assessed by optical pedobarograph
Pain score | Screening
  Assessed by patient completed Manchester foot pain and disability index

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Gusenoff, MD, Principal Investigator — University of Pittsburgh Department of Plastic Surgery; Connor Davenport, BS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Department of Plastic Surgury, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowling FL, Metcalfe SA, Wu S, Boulton AJ, Armstrong DG. Liquid silicone to mitigate plantar pedal pressure: a literature review. J Diabetes Sci Technol. 2010 Jul 1;4(4):846-52. doi: 10.1177/193229681000400412. PMID 20663447
- [Background] Abouaesha F, van Schie CH, Griffths GD, Young RJ, Boulton AJ. Plantar tissue thickness is related to peak plantar pressure in the high-risk diabetic foot. Diabetes Care. 2001 Jul;24(7):1270-4. doi: 10.2337/diacare.24.7.1270. PMID 11423514
- [Background] Abouaesha F, van Schie CH, Armstrong DG, Boulton AJ. Plantar soft-tissue thickness predicts high peak plantar pressure in the diabetic foot. J Am Podiatr Med Assoc. 2004 Jan-Feb;94(1):39-42. doi: 10.7547/87507315-94-1-39. PMID 14729989
- [Background] van Schie CH, Whalley A, Vileikyte L, Wignall T, Hollis S, Boulton AJ. Efficacy of injected liquid silicone in the diabetic foot to reduce risk factors for ulceration: a randomized double-blind placebo-controlled trial. Diabetes Care. 2000 May;23(5):634-8. doi: 10.2337/diacare.23.5.634. PMID 10834422
- [Background] 5. Van Schie CHM, Whalley A, Vileikyte L, Boulton AJM (2002) Efficacy of injected liquid silicone is related to peak plantar foot pressures in the neuropathic diabetic foot. Wounds 14:26-30
- [Background] Chairman EL. Restoration of the plantar fat pad with autolipotransplantation. J Foot Ankle Surg. 1994 Jul-Aug;33(4):373-9. PMID 7951190
- [Background] Menz HB, Tiedemann A, Kwan MM, Plumb K, Lord SR. Foot pain in community-dwelling older people: an evaluation of the Manchester Foot Pain and Disability Index. Rheumatology (Oxford). 2006 Jul;45(7):863-7. doi: 10.1093/rheumatology/kel002. Epub 2006 Jan 31. PMID 16449369
- [Background] Waldecker U. Plantar fat pad atrophy: a cause of metatarsalgia? J Foot Ankle Surg. 2001 Jan-Feb;40(1):21-7. doi: 10.1016/s1067-2516(01)80037-5. PMID 11202764